CLINICAL TRIAL: NCT04658810
Title: Assessment of Post-traumatic Stress Disorder (PTSD) in Patients Monitored for Cytomegalovirus (CMV) Seroconversion During Pregnancy, Without Ultrasound Signs or With Non-serious Ultrasound Signs of Maternal-fetal CMV Infection.
Brief Title: Assessment of Post-traumatic Stress Disorder (PTSD) in Patients Monitored for Cytomegalovirus (CMV) Seroconversion During Pregnancy,
Acronym: PTSD CMV
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1014
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Mothers; Cytomegalovirus Infections; Pregnancy Related
Keywords: CMV; Pregnancy; PTSD
MeSH Terms: conditions — Cytomegalovirus Infections; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of post-traumatic stress disorder using the Perinatal Post-traumatic Stress Disorder) — Patients identified as women with cytomegalovirus (CMV) seroconversion during pregnancy will be called on the phoned and ask to participate to the study and to answer the Perinatal Post-traumatic Stress Disorder

SUMMARY:
Reports of maternal seroconversion to CMV during pregnancy can be extremely stressful. This virus is little known to the general public and searching for information on the Internet quickly leads to a consultation of a site mentioning the risk of severe psychomotor retardation in the event of prenatal cytomegalovirus infection.

The psychological repercussions in the event of prenatal CMV infection with criteria of severity, leading or not to a request for IMG, is undeniable, but no study has investigated the consequences of seroconversion to CMV without transmission of the virus to the patient fetus, or in the case of transmission without criteria of seriousness, on the patient's experience during and after her pregnancy. Such a study would, if necessary, improve the care and support of these future mothers

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Referred to the 3 DAN centers with maternal seroconversion to CMV during their pregnancy, confirmed, with or without confirmed prenatal transmission.
* Presence of ultrasound signs without criteria of seriousness if the materno-fetal infection is proven.
* Support between January 1, 2008 and December 31, 2020.
* No opposition from patient

Exclusion Criteria:

* Reversed or anteconceptional CMV seroconversion
* Concomitant infection with another infectious agent and suspected cross-reaction
* Multiple pregnancy
* Ultrasound and / or MRI severity criteria
* Medical termination of pregnancy
* Fetal death in utero
* Birth <32 weeks and / or birth weight <1500 grams (birth criteria in maternity level IIA)
* Intercurrent event that may be the cause of an abnormality in psychomotor development
* Patients protected by justice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Assessment of post-traumatic stress disorder using the Perinatal Post-traumatic Stress Disorder)
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-05-02 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
PTSD evaluation | Through study completion, 3 months
  Assessment of post-traumatic stress disorder using the Perinatal Post-traumatic Stress Disorder scale (PPQ questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Fichez, Principal Investigator — service de Gynécologie-Obstétrique, Hôpital de la Croix Rousse
Locations (2):
- France (2):
  - Service de Gynécologie Obstétrique, Hôpital Mère Enfant, Lyon
  - Service de Gynécologie Obstétrique, Hôpital Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No